CLINICAL TRIAL: NCT00534365
Title: A Randomized Trial Comparing Tension-free Vaginal Tape (TVT) to the TVT-SECUR for the Surgical Treatment of Stress Urinary Incontinence
Brief Title: Study Comparing TVT With TVT-SECUR for the Treatment of Stress Urinary Incontinence
Acronym: SECURiTy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Good Samaritan Hospital, Ohio (Other); Greater Baltimore Medical Center (Other); Medstar Health Research Institute (Other); Duke University (Other); Foundation for Female Health Awareness (Other); Women and Infants Hospital of Rhode Island (Other); Main Line Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFHA 07-01
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; sling procedures; tension-free vaginal tape
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Tension-free vaginal tape procedure (TVT)
  Interventions: Device: tension-free vaginal tape
- 2 (Active Comparator): TVT-SECUR device
  Interventions: Device: TVT-SECUR device

INTERVENTIONS:
Device: tension-free vaginal tape — Retropubic mid-urethral sling
  Other Names: TVT
  Arms: 1
Device: TVT-SECUR device — Mid-urethral mini-sling
  Arms: 2

SUMMARY:
The purpoe of this study is to compare the safety and efficacy of the tension-free vaginal tape procedure (TVT) to the TVT-SECUR procedure in the treatment of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence symptoms
* Urodynamic stress incontinence confirmed with multichannel urodynamic testing
* Age of at least 21 years
* Desires surgical correction of stress urinary incontinence

Exclusion Criteria:

* Post-void residual volume >100cc
* Detrusor overactivity on preoperative multichannel urodynamic testing
* History of previous synthetic, biologic or fascial sub-urethral sling
* Desires future childbearing
* History of bleeding diathesis or current anti-coagulation therapy
* Current genitourinary fistula or urethral diverticulum
* Reversible cause of incontinence (i.e. drug effect)
* Contraindication to surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Barber, MD, MHS, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (7):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Main Line Health, Paoli, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island

REFERENCES:
- [Result] Barber MD, Weidner AC, Sokol AI, Amundsen CL, Jelovsek JE, Karram MM, Ellerkmann M, Rardin CR, Iglesia CB, Toglia M; Foundation for Female Health Awareness Research Network. Single-incision mini-sling compared with tension-free vaginal tape for the treatment of stress urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2012 Feb;119(2 Pt 1):328-37. doi: 10.1097/AOG.0b013e318242a849. PMID 22270285
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 281 patients were enrolled. Of these, 18 patients withdrew prior to randomization (including for the following reasons- cancelled surgery (6), did not meet inclusion criteria (4), declined further participation (8)).
Groups:
- TVT Procedure: Tension-free vaginal tape procedure (TVT)
  tension-free vaginal tape: Retropubic mid-urethral sling
- TVT-SECUR Mini Sling Procedure: TVT-SECUR device
  TVT-SECUR device: Mid-urethral mini-sling
Period: Overall Study
Arm/Group | TVT Procedure | TVT-SECUR Mini Sling Procedure
Started | 127 | 136
Received Procedure | 127 | 129 (7 patients excluded due to receipt of sling other than mini-sling)
Any Follow up | 126 | 135
Follow up at 12 Months or More | 119 | 128
Included in Intent to Treat Analysis | 127 | 136
Completed (Included in per protocol) | 127 | 129
Not Completed | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TVT Procedure | TVT-SECUR Mini Sling Procedure | Total
Number analyzed (Participants) | 127 | 136 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.3) | 54.6 (10.5) | 54.6 (11.0)
Sex/Gender, Customized [Number; unit: participants]
  Female | 127 | 136 | 263
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 120 | 118 | 238
  African American | 4 | 12 | 16
  Other | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 127 | 136 | 263
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (5.7) | 29.6 (6.4) | 29.8 (6)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Cure of Urinary Incontinence at 12 Months After Surgery
Description: Composite outcome defined as absence of urinary incontinence as indicated by the Incontinence Severity Index score of 0 and the absence of any additional surgical or nonsurgical treatment of stress urinary incontinence (SUI) after the index surgery.
Time Frame: 12 months
Population: Analysis based on per protocol enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | TVT Procedure | TVT-SECUR Mini Sling Procedure
Number analyzed (Participants) | 127 | 129
Participants | 77 | 72
Statistical Analysis 1: Comparison: TVT Procedure vs TVT-SECUR Mini Sling Procedure; Test type: Non-Inferiority or Equivalence — We chose a non-inferiority margin of 12% based on previously published multicenter trial of mid-urethral slings. Assuming subjective cure rate for TVT of 82%, 127 individuals in each group will provide 80% to reject the null hypothesis that the true difference in cure rates between the two procedures is less than or equal to 2% using a two group large sample normal approximation test of proportions with a one sided 0.05 significance level; p = 0.43, Regression, Logistic

2. Secondary Outcome: Post Operative Complications at 6 Week or Less
Time Frame: 6 week
Measure: Number; unit: participants
Arm/Group | TVT-SECUR Mini Sling Procedure | TVT Procedure
Number analyzed (Participants) | 136 | 127
participants
  Post opInfection requiring antibiotics | 5 | 6
  Urinary tract infection | 9 | 9
  Cardiac or MI | 0 | 0
  Neurologic | 0 | 0
  Pulmonary | 0 | 1
  Ileus or small bowel obstruction | 0 | 0
  Pelvic abscess | 0 | 0
  Blood transfusion | 1 | 0
  Venous thromboembolism | 1 | 0
  Return to operating room | 0 | 1
  Hospital readmissions | 2 | 2
  Emergency room evaluations | 6 | 5
  Unplanned clinic visits | 24 | 20

3. Secondary Outcome: Long Term Complications > 6 Weeks
Time Frame: 6 weeks-12 months
Measure: Number; unit: participants
Arm/Group | TVT-SECUR Mini Sling Procedure | TVT Procedure
Number analyzed (Participants) | 136 | 127
participants
  Infection requiring antibiotics | 0 | 0
  Cardiac or myocardial infection | 0 | 0
  Neurologic | 0 | 1
  Pulmonary | 0 | 0
  Ileu or small bowel obstruction | 0 | 0
  Mesh exposure | 0 | 1
  Leg pain or difficulty ambulatig | 1 | 0
  Fistula | 0 | 0

4. Secondary Outcome: Patient Global Impression Improvement
Time Frame: 12 months
Population: Please note that no all participants conducted the global improvement scale survey due to loss to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | TVT-SECUR Mini Sling Procedure | TVT Procedure
Number analyzed (Participants) | 109 | 105
Participants
  Very much better | 63 | 67
  Much better | 24 | 24
  Somewhat better | 11 | 9
  No different | 3 | 1
  Somewhat worse | 3 | 3
  Much worse | 2 | 0
  Very much worse | 3 | 1
Statistical Analysis 1: Comparison: TVT-SECUR Mini Sling Procedure vs TVT Procedure; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

5. Secondary Outcome: Incontinence Severity Index Score
Description: The incontinence severity index comprises the following two questions. How often do you experience urine leakage (0=never, 1=less than once a month, 2=one or several times a month, 3=one or several times a week, 4=every day and/or night)? How much urine do you lose each time (1=drops or little, 2=more)? The total score is the score for the first question multiplied by the score for the second question (0=dry, 1-2=slight, 3-4=moderate, 6-8=severe).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TVT-SECUR Mini Sling Procedure | TVT Procedure
Number analyzed (Participants) | 134 | 126
units on a scale | 2.2 (2.7) | 1.5 (1.9)
Statistical Analysis 1: Comparison: TVT-SECUR Mini Sling Procedure vs TVT Procedure; Test type: Superiority or Other; p = 0.015, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Intraoperative complications at time of surgery
Arm/Group | TVT-SECUR Mini Sling Procedure | TVT Procedure
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/127
Other Adverse Events (participants affected / at risk) | 6/136 | 8/127
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVT-SECUR Mini Sling Procedure (N=136) | TVT Procedure (N=127)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Blood transfusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ureteral injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Bowel injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No